CLINICAL TRIAL: NCT03162341
Title: Study of the Correlation Between UltraSonography and Dual-Energy Computed Tomography Assessment of Urate Deposit in Urate Lowering Therapy Initiators
Brief Title: Study of the Correlation Between UltraSonography and Dual-Energy Computed Tomography Assessment of Urate Deposit
Acronym: GOUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Collaborators: Horizon Pharma Rheumatology LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0056
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Gout
Keywords: Dual-Energy Computed Tomography; UltraSonography; Gout; Urate deposition
MeSH Terms: conditions — Gout | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UltraSonography and DECT (Experimental): UltraSonography and DECT will be used in patient monitoring after 6, 12 and 24 months of treatment in order to evaluate the correlation between the 2 explorations for the measurement in tophus volume change.
  Those are interventions that are not part of the standard care of the patients.
  Interventions: Procedure: ultrasonography; Procedure: DECT

INTERVENTIONS:
Procedure: ultrasonography — The tophus volume will be assess using ultrasonography.
Procedure: DECT — The tophus volume will be assess using dual-energy computed tomography (DECT).
  Other Names: dual-energy computed tomography

SUMMARY:
The objective of this research is to evaluate the correlation between DECT and US explorations performed in a routine clinical setting for the measurement of change in tophus size in gout patients after 24 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of gout based on the ACR/EULAR 2015 criteria
* uricemia ≥6 mg/dL
* warranted introduction of urate-lowering therapy according to the ACR 2012 or EULAR 2016 criteria
* signature of the informed consent
* social insurance affiliation

Exclusion Criteria:

* pregnancy or breastfeeding
* patient under legal guardianship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Correlation between US and DECT measurement of change in tophus volume | after 24 months of treatment
  Spearman rank correlation between the change in tophus volume after 24 months of treatment measured by ultrasonography or by DECT.

SECONDARY OUTCOMES:
Correlation between US and DECT measurement of change in tophus volume | after 6 months, 12 months and 24 months of treatment
  Spearman rank correlation between the change in tophus volume after 6, 12 and 24 months of treatment measured by ultrasonography or by DECT.
Change of DECT urate score | after 6 months, 12 months and 24 months of treatment
  Change from baseline after 6, 12 and 24 months of treatment in DECT urate score
Link between the change of DECT urate score and the persistence of the double contour sign | after 6 months, 12 months and 24 months of treatment
  During ultrasonography, a double contour of the articulation can be visible. This outcome will compare the change in the DECT urate score between the patients for who the double contour stay visible and those for who it disapear.
  This outcome register if this double contour stay visible.
Correlation between the change of DECT urate score and the change in serum uric acid levels | after 6 months, 12 months and 24 months of treatment
  The Spearman correlation between the change from baseline of the DECT urate score and the serum uric acid levels will be computed for each time point.
Correlation between the change of DECT urate score and the number of gout attacks | after 6 months, 12 months and 24 months of treatment
  The Spearman correlation between the change from baseline of the DECT urate score and the number of gout attack will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Pascart, MD, Study Director — Hospital Group of the Catholic Institute of Lille; Sébastien Ottaviani, MD, Principal Investigator — Bichat Hospital of Paris; Pascal Richette, MD PhD, Principal Investigator — Lariboisiere Hospital of Paris
Locations (3):
- France (3):
  - Hospital Group of the Catholic Institute, Lomme
  - Bichat Hospital, Paris
  - Lariboisière Hospital, Paris

IPD SHARING:
Plan to Share IPD: Undecided